CLINICAL TRIAL: NCT01160601
Title: A Randomized, Open-Label, Phase 2 Trial of Paclitaxel/Carboplatin With or Without Bavituximab in Patients With Previously Untreated Locally Advanced or Metastatic Non-Squamous Non Small-Cell Lung Cancer
Brief Title: Study of Paclitaxel/Carboplatin With or Without Bavituximab in Previously Untreated Non Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 1001
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
Keywords: NSCLC; lung cancer; non small cell lung cancer; bavituximab; monoclonal antibody
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — CP protocol; bavituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- paclitaxel/carboplatin plus bavituximab (Experimental): Patients will receive paclitaxel (200 mg/m2) and carboplatin (target area under the concentration-time curve [AUC] 6) on Day 1 of each 21 day cycle for up to 6 cycles, in combination with 3 mg/kg bavituximab administered weekly.
  Interventions: Drug: Paclitaxel / Carboplatin; Drug: bavituximab
- paclitaxel/carboplatin (Active Comparator): Patients will receive paclitaxel (200 mg/m2) and carboplatin (target area under the concentration-time curve [AUC] 6) on Day 1 of each 21 day cycle for up to 6 cycles.
  Interventions: Drug: Paclitaxel / Carboplatin

INTERVENTIONS:
Drug: Paclitaxel / Carboplatin — Patients will receive commercially available paclitaxel (200 mg/m2) and carboplatin (target area under the concentration-time curve [AUC] 6) on Day 1 of each 21 day cycle for up to 6 cycles.
Drug: bavituximab — Patients will receive 3 mg/kg bavituximab, administered weekly until progression or toxicity.
  Arms: paclitaxel/carboplatin plus bavituximab

SUMMARY:
This is a randomized, open-label, multicenter, phase 2 study comparing Paclitaxel/Carboplatin with or without bavituximab in patients that have previously untreated locally advanced or metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Key Inclusion Criteria:

* Adults over 18 years of age with a life expectancy of at least 3 months.
* Histologically or cytologically confirmed stage IIIB or stage IV non-squamous NSCLC that has not been previously treated with systemic chemotherapy.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST, Version 1.1).
* Adequate hematologic, renal and hepatic function.
* PT / INR ≤ 1.5 × ULN, aPTT ≤ 1.5 × ULN and D-dimer ≤ 3 × ULN.

Key Exclusion Criteria:

* Squamous cell, small cell, or mixed histology.
* Known history of bleeding diathesis or coagulopathy.
* Cavitary tumors or tumors abutting large blood vessels.
* Bleeding: Clinically significant bleeding, such as gross hematuria, GI bleeding and hemoptysis, within 12 months of Screening.
* Venous thromboembolic events (e.g., deep vein thrombosis or pulmonary thromboembolism) within 6 months of Screening.
* Ongoing therapy with oral or parenteral anticoagulants.
* Concurrent estrogens, anti-estrogens or progesterone compounds.
* Grade 2 or higher peripheral neuropathy.
* Radiotherapy within 2 weeks preceding Study Day 1.
* Symptomatic or clinically active brain metastases.
* Major surgery within 4 weeks of Study Day 1.
* Uncontrolled intercurrent disease (e.g., diabetes, hypertension, thyroid disease).
* Symptomatic coronary artery disease, cerebrovascular accident,transient ischemic attack, myocardial infarction, or unstable angina pectoris within 6 months of Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | Until disease progression

CONTACTS AND LOCATIONS:
Locations (40):
- United States (17):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - Baptist Clinical Research, Jonesboro, Arkansas
  - American Institute of Research, Whittier, California
  - Baptist Cancer Institute, Jacksonville, Florida
  - Community Hospital, Munster, Indiana
  - Cedar Valley Medical Specialists, PC, Waterloo, Iowa
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Presbyterian Hospital, Charlotte, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - The Christ Hospital Cancer Center Research, Cincinnati, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Hematology-Oncology of Knoxville/Mercy Medical Center, Knoxville, Tennessee
  - Delta Hematology Oncology Associates, PC, Portsmouth, Virginia
- Georgia (2):
  - JSC A.Gvamichava National Oncology Center, Tbilisi
  - Medulla Chemotherapy and Immunotherapy Clinic, Tbilisi
- India (9):
  - BiBi General Hospital & Cancer Centre, Hyderabad, Andhra Pradesh
  - Mahavir Cancer Sansthan, Patna, Bihar
  - O.P. Jindal Institute of Cancer & Research, Hisar, Haryana
  - Bangalore Institute of Oncology Specialty Centre, Bangalore, Karnataka
  - Kodlikeri Memorial Hospital, Aurangabad, Maharashtra
  - Cancer Care Clinic, Nagpur, Maharashtra
  - Shatabdi Superspecialty Hospital, Nashik, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - SMS Medical College Hospital, Jaipur, Rajasthan
- Russia (7):
  - State Institution of Healthcare "Pyatigorsk Oncology Dispensary", Pyatigorsk, Stavropol Territory
  - State Institution of Healthcare of Yaroslavl Region "Regional Clinical Oncology Hospital", Yaroslavl, Yaroslavl Oblast
  - State Medical Preventive Institution "Chelyabinsk Regional Clinical Oncology", Chelyabinsk
  - State Institution of Healthcare " Ivanovo Regional Oncology Dispensary ", Ivanovo
  - Institution of Russian Academy of Medical Science "Russian Oncology Scientific Centre named after N. N. Blokhina RAMN", Moscow
  - State Educational Institution of Higher Professional Education "Saint-Petersburg State Medical University named after academician I.P. Pavlov of Federal Agency of Healthcare and Social Development", Saint Petersburg
  - State Institution of Healthcare "Tula Regional Oncology Dispensary", Tula
- Ukraine (5):
  - City multi-field clinical hospital # 4, Department of chemotherapy; Dnipropetrovsk State Medical Academy, Chair of Oncology and Medical Radiology;, Dnipropetrovsk
  - Municipal Clinical Medical and Prophylactic Institution "Donetsk Regional Antineoplastic Center", onco-chemotherapy department #1, Donetsk
  - State Institution "Institute of Medical Radiology named after S.P. Grygoryev of AMS of Ukraine", department of chemotherapy, Kharkiv
  - Kyiv City Oncology Hospital, Thoracal Department, Kyiv
  - Uzhgorod Central City Clinical Hospital, City Oncology Center, Uzhhorod